CLINICAL TRIAL: NCT02102815
Title: Efficacy of Preoperative Intravenous Dexamethasone in Controlling Postoperative Pain After Primary Total Knee Arthroplasty: A Randomized Double-blinded Controlled Trial
Brief Title: Efficacy of Preoperative Intravenous Dexamethasone in Primary Total Knee Arthroplasty
Acronym: TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, Orthopaedics department, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OrthoTU06
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Pain
Keywords: total knee arthroplasty; pain control; dexamethasone; steroids
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Experimental): Preoperative dexamethasone 0.15mg/Kg mixed with NSS to 50 mL IV slowly push over 5 minutes
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Preoperative intravenous normal saline 50 mL slowly push over 5 minutes
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 0.15mg/kg mixed with NSS up to 50 mL IV slowly push over 5 minutes
  Arms: Dexamethasone
Drug: Normal saline — NSS 50 mL IV slowly push over 5 minutes
  Arms: Placebo

SUMMARY:
To determine efficacy of preoperative IV dexamethasone for postoperative pain control after TKA.

DETAILED DESCRIPTION:
Preoperative intravenous over 0.1 mg/kg of dexamethasone could be reduced pain after primary TKA.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee who undergoing unilateral primary total knee arthroplasty
* 50-85 years old
* ASA class 1-3

Exclusion Criteria:

* Unable to perform spinal anaesthesia
* History of drug allergies: steroids
* Renal impairment (CrCl <30 mL/min)
* Liver impairment
* Cognitive function disorders
* Poor controlled DM (HA1C > 7.5)
* Morning DTX at operative day > 180 mg%
* Received corticosteroids within 3 months before surgery

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
post-operative pain | 48 hours
  measured with VAS for pain, drugs for relief pain

SECONDARY OUTCOMES:
Functional knee score | 3 month
  measured with WOMAC, KSS
post-operative nausea and vomiting | 48 hours
  measured with amount of nausea/vomiting and drugs requiring for fixed its.
complication of preoperative dexamethasone | 2 weeks
  measured with wound complication, blood sugar level
inflammatory level | 48 hours
  CRP level

OTHER OUTCOMES:
Knee range of motion | 3 months
  measuring range of motion with goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Supakit Kanitnate, M.D., Principal Investigator — Orthopaedics department, Thammasat University
Locations (1):
- Orthopaedic department, Faculty of medicine, Thammasat university, Klongluang, Changwat Pathum Thani, Thailand